CLINICAL TRIAL: NCT00885937
Title: Single-blind, Randomized, Controlled, Single Center Trial to Evaluate the Skin Irritation Potential of a New Topical Formulation by Means of an Occlusive Patch Test in Healthy Subjects.
Brief Title: Comparative Safety Study of New Sinecort Formulation Versus Positive Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 13941; 2008-008138-36 (EudraCT Number); Sinecort (Other: Company Internal)
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Dexpanthenol; Safety,; New formulation; Topical administration
MeSH Terms: interventions — dexpanthenol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Dexpanthenol (Sinecort, BAY81-2996)
- Arm 2 (Active Comparator)
  Interventions: Drug: Positive control, Na-laurylsulfat-solution
- Arm 3 (Placebo Comparator)
  Interventions: Device: Untreated skin under application chamber

INTERVENTIONS:
Drug: Dexpanthenol (Sinecort, BAY81-2996) — 1 squeeze of Sinecort cream sufficient to cover the area of the application chamber, (=50 mikro liter)
  Arms: Arm 1
Drug: Positive control, Na-laurylsulfat-solution — 50 mikro liter of 0.5 % Sodium-laurylsulfate-solution
  Arms: Arm 2
Device: Untreated skin under application chamber — Application of treatment chamber as in arm 1 and arm 2 on untreated skin
  Arms: Arm 3

SUMMARY:
The study is focused to prove a favorable safety profile of the new formulation.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Skin type I, II, or III according to Fitzpatrick
* Subjects of childbearing potential must use an acceptable method of contraception. Hormonal or oral contraceptive drugs, intra-uterine devices (IUD) and abstinence are considered acceptable methods of contraception.

Exclusion Criteria:

* Clinical history suggestive of intolerance, allergies or idiosyncrasies to one of the products or the ingredients of the products including the patch.
* Known skin allergies.
* Dermatologic diseases that might interfere with the evaluation of test site reaction.
* Other(s), considered as important by the investigator (e.g. multiple birth marks in the test area, important hair growth in the test area, pigmented or extremely suntanned skin impairing visual assessment, tattoos in the test area.
* Topical use of any cosmetic preparation on the test areas within 5 days prior to Day 1 (Start of Treatment) or during the trial
* Within 3 weeks prior to Day 1 and during the entire trial. Any systemic or topical medication likely to interfere with the trial purposes: e.g. immune-modulating therapy (e.g. corticosteroids, cytotoxics or immunosuppressants) and any dermatological medication (drug or medical device.
* Within 1 week prior to Day 1 and during the entire trial any medication with common effects on the perfusion of skin vessels (e.g. vasodilators or vasoconstrictors, ß-receptor blocking drugs, antihistamines) should not be used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Irritation rate | After 21 applications

SECONDARY OUTCOMES:
Irritation potential | After 21 applications

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Münster, North Rhine-Westphalia, Germany